CLINICAL TRIAL: NCT03580603
Title: The Effect of Data Visualization on Provider Knowledge of Culture Sensitivity Results
Brief Title: Clinical Decision Support Tools for Antibiotic Prescribing
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Beth Israel Deaconess Medical Center (Other)
Responsible Party: Principal Investigator, Steven Horng, MD, Principal Investigator, Beth Israel Deaconess Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 2017P000432; 2017P000432 (Other: Committee on Clinical Investigations Beth Israel Deaconess Medical Center)
Record Dates: First submitted 2018-04-09; First posted 2018-07-09 (Actual); Last update posted 2021-05-06 (Actual); Status verified 2021-05

CONDITIONS: Infectious Disease
MeSH Terms: conditions — Communicable Diseases

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Antibiotic visualization tool (Experimental): Provider will answer microbiological sensitivity questions using a new antibiotic visualization tool.
  Interventions: Other: Visualization tool
- Standard practice (No Intervention): Provider will answer microbiological sensitivity questions using standard medical record tools.

INTERVENTIONS:
Other: Visualization tool — Visual representation of past microbiological culture data
  Arms: Antibiotic visualization tool

SUMMARY:
The goal of this study is to assess the utility of a data visualization tool for providers' understanding patients' past microbiological culture sensitivities. Providers that are ordering antibiotics for patients with previous culture data in the medical record will be asked to answer questions regarding past sensitivity results. They will be randomized to either using the visualization tool before answering the questions or using the standard medical record tools. They will then be surveyed about their decision-making, knowledge, and the usefulness of the tool.

ELIGIBILITY:
Inclusion Criteria:

* provider is caring for a patient with a previous positive urine or blood cultures
* provider is caring for a patient currently in a clinical location being investigated
* provider is caring for a patient with orders placed for an intravenous, intramuscular, oral antibiotics

Exclusion Criteria:

* the patient has already received the antibiotic by the time of the intervention
* the antibiotic has been cancelled by the time of intervention
* the research assistant is unable to reach the ordering provider before the visit is completed
* participation by the clinician in the study would impede clinical care
* age < 18

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 273 (Actual)
Dates: Start 2018-03-05 (Actual); Primary Completion 2018-09-30 (Actual); Study Completion 2018-09-30 (Actual)

PRIMARY OUTCOMES:
Provider knowledge | To be assessed at the time of patient enrollment, up to one day after the initial antibiotic is ordered.
  Provider knowledge of patients' previous culture sensitivity results as determined by the proportion of correct answers on a questionnaire:
  Do you think this patient has had previous resistance to each of these antibiotics at BIDMC (Beth Israel Deaconess Medical Center)?
  [List of the top 4 antibiotic classes to which resistance is seen at BIDMC that the patient has previously had tested for antibiotic sensitivities]
  Yes (previous organisms resistant or with intermediate resistance)
  No (no previous resistance noted)

SECONDARY OUTCOMES:
Post-intervention survey | To be assessed at the time of patient enrollment, up to one day after the initial antibiotic is ordered.
  Providers will be asked survey questions regarding their decision-making and the usability and usefulness of the tool using a 5 point Likert scale:
  I understand the previous culture data for this patient (Strongly disagree) 1 2 3 4 5 (Strongly agree)
  I feel like I made an informed antibiotic choice (Strongly disagree) 1 2 3 4 5 (Strongly agree)
  The tool provided new information that you were not previously aware of (Strongly disagree) 1 2 3 4 5 (Strongly agree)
  The tool enabled you to more quickly understand this patient's microbiological data (Strongly disagree) 1 2 3 4 5 (Strongly agree)
  The tool was easy to use (Strongly disagree) 1 2 3 4 5 (Strongly agree)
Antibiotic order changes | To be assessed at the time of patient enrollment + 1 day
  Antibiotic orders that are not complete by the time of the intervention will be monitored for any cancellation or change in orders
Final culture results | To be assessed at the time of patient enrollment + 1 week
  Final culture results drawn from that visit will be compared to antibiotic orders for effectiveness

CONTACTS AND LOCATIONS:
Overall Officials: Steven Horng, MD, Principal Investigator — Beth Israel Deaconess Medical Center
Locations (1):
- Beth Israel Deaconess Medical Center, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: Undecided